CLINICAL TRIAL: NCT01756508
Title: Study of Eculizumab for Prevention and Treatment Reperfusion Injury in Kidney Transplantation.
Brief Title: Eculizumab for Prevention and Treatment of Kidney Graft Reperfusion Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Russian Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Michael Kaabak, professor, Russian Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Eculizumab for reperfusion
Record Dates: First submitted 2012-12-20; First posted 2012-12-27 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: End-Stage Renal Disease; Kidney Failure; Graft Reperfusion Injury
Keywords: eculizumab; kidney transplantation; reperfusion; rejection; infection
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency; Rejection, Psychology; Infections | interventions — eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- eculizumab (Experimental): Eculizumab 1200 mg/m2 will be administered once, 1 hour before graft reperfusion
  Interventions: Drug: eculizumab
- control (No Intervention): No intervention will be applied instead eculizumab infusion

INTERVENTIONS:
Drug: eculizumab — Eculizumab 1200 mg/m2 will be administered once, 1 hour before graft reperfusion
  Other Names: Soliris
  Arms: eculizumab

SUMMARY:
Study of eculizumab ability to correct the reperfusion injury of the kidney allograft.

DETAILED DESCRIPTION:
Based on experimental data and supportive observations in humans associating complement gene upregulation with ischemic reperfusion injury, it is hypothesized that C5 cleavage is a key step in the pathogenesis of ischemic reperfusion injury following transplantation. It was further hypothesized that eculizumab, antibody that blocks C5 cleavage in humans will be an effective prophylactic agent to prevent ischemic reperfusion injury in high risk recipients. For testing this hypothesis, this study is a pilot prospective study to test the efficacy of eculizumab in preventing the development of reperfusion injury and contribute graft survival.

ELIGIBILITY:
Inclusion Criteria:

1. age 1-80
2. weight - >6 kg
3. male or female
4. recipient of first kidney graft either from standard criteria deceased or live donor
5. end stage renal disease or congenital nephrotic syndrome -

Exclusion Criteria:

1. Blood group (ABO) incompatible transplantation
2. presence of donor-specific anti-human leukocyte antigen (HLA) antibodies
3. multiorgan transplantation
4. previous transplant
5. patients infected with HIV, hepatitis C virus (HCV) or hepatitis B virus (HBV)
6. patients with haemolytic-uraemic syndrome (HUS) -

Ages: 12 Months to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2012-09-01 (Actual); Primary Completion 2017-04-15 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
speed of the graft warming | at the time of engraftment
  The speed of the graft surface warming in the range 15-20°C is accessed on the the infrared video record, taken during graft reperfusion by Nec Thermo Tracer.

SECONDARY OUTCOMES:
graft morphology changes | one year after transplantation
  Protocol biopsy will be obtained at one month and one year. Progression of allograft nephropathy will be compared between groups.
One-year graft and patient survival, as well as rejection and infection rates will be calculated | one year after Tx
primary graft function | first week after Tx
  initial graft function will be accessed daily during the first week post Tx and measured as follows:
  * the rate of serum creatinine decrease expressed as percent per day, where 100% will be the creatinine on the day before;
  * intragraft blood flow by Doppler indexes (acceleration, resistance) and blood flow velocity on the three levels - main, interlobar and arcuate arteries;

CONTACTS AND LOCATIONS:
Overall Officials: Michael M Kaabak, MD, Principal Investigator — Russian Scientific Center of Surgery
Locations (1):
- Russian Scientfic Center of Surgery, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data, except for personal data like Name, Forename, and address, will be shared by request

REFERENCES:
- [Background] de Vries DK, van der Pol P, van Anken GE, van Gijlswijk DJ, Damman J, Lindeman JH, Reinders ME, Schaapherder AF, Kooten Cv. Acute but transient release of terminal complement complex after reperfusion in clinical kidney transplantation. Transplantation. 2013 Mar 27;95(6):816-20. doi: 10.1097/TP.0b013e31827e31c9. PMID 23348894
- [Background] Kaabak M, Babenko N, Shapiro R, Zokoyev A, Dymova O, Kim E. A prospective randomized, controlled trial of eculizumab to prevent ischemia-reperfusion injury in pediatric kidney transplantation. Pediatr Transplant. 2018 Mar;22(2). doi: 10.1111/petr.13129. Epub 2018 Jan 29. PMID 29377474